CLINICAL TRIAL: NCT06085118
Title: Prospective National Observatory for Cow's Milk Protein Allergy.
Brief Title: Observatory on Cow's Milk Protein Allergy
Acronym: OLAF
Status: Recruiting | Type: Observational
Sponsor: Nutricia Nutrition Clinique (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A01285-40
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Infants up to and including 8 months of age (up to 8 months and 29 days), treated for a suspected or confirmed cow protein allergy.
  Interventions: Other: Pepticate® Syneo®

INTERVENTIONS:
Other: Pepticate® Syneo® — Introduction of the nutritional treatment Pepticate® Syneo® (high protein hydrolysate), as a foodstuff for special medical purposes (product already available on the market).

SUMMARY:
The purpose of this study is to describe the symptoms and their evolution up to the age of 5 years in a population of newly diagnosed infants with a suspected or confirmed allergy to cow proteins, for whom the doctor prescribed the Pepticate® Syneo® replacement formula as soon as they were diagnosed.

The Pepticate® Syneo® product is an advanced protein hydrolyzate, food type intended for special medical purposes. This is a product already available on the market.

DETAILED DESCRIPTION:
This is a prospective, observational, descriptive, longitudinal, multicentric study aimed at describing a cohort of infants with a recently suspected or confirmed allergy to cow's milk protein, who were treated in outpatient and inpatient settings.

The recruitment of patients eligible for this observatory will be done via community medicine (private practices of pediatricians and general practitioners) as well as in hospitals throughout France.

ELIGIBILITY:
Inclusion Criteria:

* Infants up to and including 8 months (up to 8 months and 29 days).
* Initial diagnosis of allergy to cow proteins, suspected (clinical presumption) or confirmed.
* Prescription of the substitution formula Pepticate® Syneo, according to the doctor's judgement, whether the child is under mixed or weaned breastfeeding.
* Authorisation from a legal representative for the child to take part in the observatory and to collect personal information about the child and the family.
* Membership of the social security system.

Exclusion Criteria:

* Infants who have already received partial or total replacement infant formula (regardless of the type of infant formula).
* Contraindication to the use of symbiotics (short small intestine, parenteral nutrition, post-pyloric feeding, central venous catheter) due to the use of Pepticate® Syneo®.
* Diagnosis of severe cow protein allergy requiring an infant amino acid formula from the outset.
* The child's legal guardian is protected (under legal protection, or deprived of liberty by judicial or administrative decision).
* The legal representative is unable to understand the study protocol.

Max Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population of our project will be infants up to and including 8 months of age (up to 8 months and 29 days), treated for a suspected or confirmed, newly diagnosed cow protein allergy requiring, according to the investigator's judgement, an initial prescription of the Pepticate® Syneo® advanced cow protein hydrolysate infant formula.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of symptoms | 5 years
  Numbers and proportion of symptoms (cutaneous, gastrointestinal, respiratory...), and their evolution according to the different forms of cow protein allergy: immediate Immunoglobulin E mediated, delayed non-Immunoglobulin E mediated or mixed and acute food protein-induced enterocolitis syndrome.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Cabinet du Dr Phu My TRAN, Nice
  - Hôpital Trousseau - APHP, Paris